CLINICAL TRIAL: NCT04269538
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY OPEN, PLACEBO-CONTROLLED, DOSE ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS FOLLOWING SINGLE SUBCUTANEOUS DOSE OF PF-06480605 IN JAPANESE HEALTHY PARTICIPANTS
Brief Title: Evaluation of Safety, Tolerability and Pharmacokinetics of Single Dose of PF-06480605 in Japanese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telavant, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7541006
Record Dates: First submitted 2020-01-22; First posted 2020-02-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD Cohorts 1-2 Experimental Arm (Experimental): Experimental Arm Active drug 150 mg and 450 mg SC dosing
  Interventions: Drug: PF-06480605
- SAD Cohorts 1-2 Placebo Arm (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06480605 — PF-06480605 150 mg and 450 mg SC dosing
  Other Names: Cohorts 1 and 2 Active
  Arms: SAD Cohorts 1-2 Experimental Arm
Drug: Placebo — Placebo SC dosing
  Arms: SAD Cohorts 1-2 Placebo Arm

SUMMARY:
This is a Phase 1, randomized, double-blind, third-party open (ie, participant-blind, investigator-blind and sponsor-open), placebo-controlled, dose escalating clinical study to evaluate the safety, tolerability, immunogenicity, PK and PD of PF-06480605 in Japanese healthy adult participants.

DETAILED DESCRIPTION:
Approximately 16 participants are planned to be enrolled into the study. The study consists of 2 cohorts, and approximately 6 participants will be randomized to PF-06480605 and approximately 2 participants will be randomized to placebo in each cohort. Each participant will receive PF-06480605 or placebo subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 20 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Participants must have four Japanese grandparents born in Japan.
3. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, cardiac tests and laboratory tests.
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
5. Body mass index (BMI) of 17.5 to 25 kg/m2; and a total body weight >50 kg (110 lb).
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of human immunodeficiency virus (HIV) infection, hepatitis C or syphilis; positive testing for HIV, hepatitis C antibody (HCVAb) or syphilis.
3. Infection with hepatitis B (HBV) according to the following algorithm using the results of positive testing for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) and hepatitis B surface antibody (HBsAb) at screening.

   1. If all three tests are negative, the participant is eligible for study inclusion.
   2. If HBsAg is positive, the participant must be excluded from participation in the study.
   3. If HBsAg is negative, HBcAb is positive, and HBsAb is negative, the participant must be excluded from participation in the study.
   4. If HBsAg is negative, HBcAb is negative, HBsAb is positive, and prior HBV vaccination is unequivocally documented, the participant is eligible for the study and does not require hepatitis B DNA (HBVDNA) monitoring during the study.
   5. If HBsAg is negative, HBcAb is negative, HBsAb is positive, and no unequivocal documentation of prior HBV vaccination is available, the participant is required to undergo HBVDNA reflex testing:

   i. If HBVDNA is detected, the participant must be excluded from participation in the study; ii. If HBVDNA is undetectable, the participant is eligible for study inclusion. If the participant is included in the study, for subsequent visits HBVDNA testing must be performed according to the Schedule of Activities.

   f. If HBsAg is negative, HBcAb is positive, and HBsAb is positive, the participant is required to undergo HBVDNA reflex testing: i. If HBVDNA is detected, the participant must be excluded from participation in the study; ii. If HBVDNA is undetectable, the participant is eligible for study inclusion. If the participant is included in the study, for subsequent visits HBVDNA testing must be performed according to the Schedule of Activities.
4. History of allergic or anaphylactic reaction to a therapeutic drug.
5. History of recent active infections within 28 days prior to the screening visit.
6. Participants with a fever within 48 hours prior to dosing.
7. History of tuberculosis or active, latent or inadequately treated tuberculosis infection as defined by the following:

   Have evidence of untreated or inadequately treated active or latent Mycobacterium tuberculosis (TB) infection as evidenced by the following:
   1. A positive QuantiFERON TB Gold In Tube (QFT-G) test or positive or borderline T-SPOT.TB (T Spot) test performed within the 12 weeks prior to Day 1. If the laboratory reports the test as indeterminate, the test should be repeated. If the result of the repeat test is indeterminate, a purified protein derivative (PPD) test may be substituted for the QFT-G test or T-Spot test only with approval from the Pfizer Medical Monitor on a case by case basis.
   2. Chest radiograph with changes suggestive of active TB infection within 3 months prior to Screening. Chest radiograph should be performed according to local standards of care or country specific guidelines.
   3. History of either untreated or inadequately treated latent or active TB infection.

   If a participant has previously received an adequate course of therapy for either latent (9 months of isoniazid in a locale where rates of primary multi drug resistant TB infection are <5% or an acceptable alternative regimen) or active (acceptable multi drug regimen) TB infection, neither a QFT-G test, a T-Spot test, nor a PPD test need be obtained. Details of the previous course of therapy (eg, medication(s) used, dose, duration of therapy) should be documented in the source documentation.

   A chest radiograph should be obtained if not done within the 3 months prior to Screening. To be considered eligible for the study, the chest radiograph must be negative for active TB infection.

   A participant who is currently being treated for active TB infection must be excluded from the study.

   A participant who is being treated for latent TB infection can only be enrolled with confirmation of current incidence rates of multi drug resistant TB infection, documentation of an adequate treatment regimen, and prior approval of the Sponsor.
8. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
9. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product.
10. Recent exposure to live vaccines within 28 days of the screening visit.
11. Known exposure to anti-TL1A (PF-06480605) or any type of anti-TL1A therapy.
12. Previous administration with an investigational drug within 4 months (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).
13. A positive urine drug test.
14. Screening supine blood pressure (BP) >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
15. Baseline 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete left bundle branch block [LBBB], signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
16. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
17. Blood donation (excluding plasma donations and platelet donations) of approximately >=400 mL within 3 months or >=200 mL within a month prior to dosing. Additionally, approximately >=400 mL within 4 months for female participants.
18. History of sensitivity to heparin or heparin induced thrombocytopenia.
19. History of substance abuse within 12 months of the screening visit.
20. Pregnant females; breastfeeding females.
21. Males who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and until discharge from the study.
22. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
23. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events (AEs). | Day 0-114
Incidence, severity and causal relationship of treatment emergent AEs (TEAEs) and withdrawals due to treatment emergent adverse events. | Day 0-114
Incidence and magnitude of abnormal laboratory findings. | Day 0-114
Incidence of abnormal and clinically relevant changes in pulse rate | Day 0-114
  The use of an automated device for measuring pulse rate is acceptable; however, when done manually, pulse rate will be measured in the brachial/radial artery for at least 30 seconds.
Incidence of abnormal and clinically relevant changes in supine blood pressure | Day 0-114
  The use of an automated device for measuring blood pressure is acceptable; however, when done manually, pulse rate will be measured in the brachial/radial artery for at least 30 seconds.
Incidence of abnormal and clinically relevant changes in temperature | Day 0-114
  Temperature will be measured orally. No eating, drinking, or smoking is allowed for 15 minutes prior to the measurement.
Incidence of abnormal and clinically relevant changes in electrocardiogram | Day 0-114
  12-Lead electrocardiograms should be collected using an electrocardiogram machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. All scheduled ECGs should be performed after the participant has rested quietly for at least 10 minutes in a supine position.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Day 0-114
Time to reach maximum observed serum concentration (Tmax) | Day 0-114
Area under the serum concentration-time profile from time zero to 14 days (AUC14 days) | Day 0-114
Terminal elimination half-life (t1/2) | Day 0-114
Apparent volume of distribution (Vz/F) | Day 0-114
Apparent total body clearance (CL/F) | Day 0-114
Immunogenicity of PF-06480605 | Day 0-114
  Incidence of the development of anti-drug antibody (ADA) and neutralizing antibody (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Hachioji-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fukuhara K, Neelakantan S, Furihata K, Yuasa H, Shi N, Yamamoto Y, Hung KE. Japanese Phase 1 Study for Global Development of Anti-TL1A Antibody PF-06480605: A Randomized, Placebo-Controlled, Single-Ascending Dose Study. Clin Transl Sci. 2025 Mar;18(3):e70187. doi: 10.1111/cts.70187. PMID 40065559
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7541006